CLINICAL TRIAL: NCT04433455
Title: Influencing Factors of Cerebrovascular Disease and Cognition in Hemodialysis Patients: an Observational Study
Brief Title: Influencing Factors of Cerebrovascular Disease and Cognition in Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Professor, Huashan Hospital
Other Study IDs: KY2019-465
Record Dates: First submitted 2020-05-19; First posted 2020-06-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hemodialysis; Cognitive Impairment; Cerebrovascular Disorders
MeSH Terms: conditions — Cognitive Dysfunction; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this observational study, the investigators evaluate the influencing factors of cerebrovascular disease and cognition in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. maintenance hemodialysis patients who are younger than 85 years old and older than 50 years old, regardless of gender
2. dialysis vintage is greater than 3 months;

Exclusion Criteria:

1. Those with severe infection and anemia (Hb <60g / L);
2. Those with severe mental illness, metabolic diseases and immune system diseases;
3. Patients with abnormal liver function

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: maintenance hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
cerebrovascular disease | 5 years
  Magnetic resonance images will be used to determine the severity of white matter hyperintensity, using the Scheltens scale. Score 2 or more is abnormal.

SECONDARY OUTCOMES:
changes in cognitive function | 5 years
  The Mini-Mental State Examination (MMSE) will be used to assess the changes in cognitive function.The MMSE has a maximum score of 30 points. The scores are generally grouped as follows:
  25-30 points: normal cognition 21-24 points: mild dementia 10-20 points: moderate dementia 9 points or lower: severe dementiaThe Mini-Mental State Examination (MMSE) will be used to assess the changes in cognitive function.The MMSE has a maximum score of 30 points. The scores are generally grouped as follows: 25-30 points: normal cognition 21-24 points: mild dementia 10-20 points: moderate dementia 9 points or lower: severe dementia

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China